CLINICAL TRIAL: NCT00543374
Title: A Phase III, Multicenter, Placebo-controlled, Randomized, Double-blind Durability and Retreatment Study to Evaluate the Safety and Efficacy of PROCHYMAL® (ex Vivo Cultured Adult Human Mesenchymal Stem Cells) Intravenous Infusion for the Maintenance and Re-induction of Clinical Benefit and Remission in Subjects Experiencing Treatment-refractory Moderate-to-severe Crohn's Disease
Brief Title: Extended Evaluation of PROCHYMAL® Adult Human Stem Cells for Treatment-Resistant Moderate-to-Severe Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mesoblast, Inc. (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRD 610
Record Dates: First submitted 2007-10-11; First posted 2007-10-15 (Estimated); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PROCHYMAL Low dose (Active Comparator): Low dose (total of 600 million cells)
  Interventions: Drug: PROCHYMAL adult human mesenchymal stem cells
- PROCHYMAL High dose (Active Comparator): High dose (total of 1200 cells)
  Interventions: Drug: PROCHYMAL adult human mesenchymal stem cells

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: PROCHYMAL adult human mesenchymal stem cells — intravenous infusion four times over two weeks; possibly repeated once
  Arms: PROCHYMAL High dose; PROCHYMAL Low dose

SUMMARY:
Protocol 610 is enrolling subjects who successfully achieved clinical benefit (reduction in Crohn's Disease Activity Index (CDAI) of at least 100 points) in Protocol 603. Protocol 610 is evaluating the length of initial effect of PROCHYMAL® adult human mesenchymal stem cells and the ability of these cells to successfully re-induce clinical benefit.

DETAILED DESCRIPTION:
A significant number of individuals with Crohn's disease do not find relief with existing steroidal, immunosuppressive, or biologic therapies, and are forced to seek surgery or other drastic measures for treatment.

PROCHYMAL® adult human stem cells are manufactured from healthy, volunteer donors, extensively tested, and are stored to be available as needed. Human and animal studies have shown that the cells do not require any donor-recipient matching. The cells may have both immunosuppressive and healing benefits in Crohn's disease. The cells naturally migrate specifically to sites of inflammation, so their effects are believed to be local and self-limiting rather than systemic.

Protocol 610 is an extension study offered only to those subjects who successfully achieved clinical benefit (reduction of CDAI of at least 100 points) in Protocol 603.

ELIGIBILITY:
Inclusion Criteria:

* Participation in Osiris Protocol 603, with drop of at least 100 points in CDAI at Day 28

Exclusion Criteria:

* Substance abuse
* Failure to receive full dose of all interventions in Protocol 603

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-09-17 (Actual); Primary Completion 2009-07 (Actual); Study Completion 2011-04-28 (Actual)

PRIMARY OUTCOMES:
Duration of clinical benefit (Crohn's disease activity index) | 6 months
Re-induction of clinical benefit (Crohn's disease activity index) | 6 months

SECONDARY OUTCOMES:
Improvement in quality of life (Inflammatory Bowel Disease Questionnaire [IBDQ] instrument) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahboob Rahman, MD, Study Director — Mesoblast, Inc.
Locations (58):
- United States (53):
  - Advanced Clinical Research Institute, Anaheim, California
  - Veteran's Administration Medical Center (does not require vet status), Long Beach, California
  - University of Southern California University Hospital, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Western States Clinical Research, Wheat Ridge, Colorado
  - Gastroenterology Center of Connecticut, Hamden, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Venture Research Institute, Miami, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Topeka, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Gulf Coast Research, Baton Rouge, Louisiana
  - National Institutes of Health, Bethesda, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Center for Clinical Studies, Dearborn, Michigan
  - Center for Digestive Health, Troy, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - St Louis Center for Clinical Studies, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Gastroenterology Research Associates, Cedar Knolls, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Rochester Institute for Digestive Diseases, Rochester, New York
  - Rochester General Hospital, Rochester, New York
  - University Hospital and Medical Center, Stony Brook, New York
  - Charlotte Gastroenterology and Hepatology, Charlotte, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Dayton Science Institute, Dayton, Ohio
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Allegheney Center for Digestive Health, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Gastroenterology Center of the Midsouth, Germantown, Tennessee
  - Nashville GI Specialists, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - University of Vermont, Burlington, Vermont
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
  - McGuire Research Institute, Richmond, Virginia
  - Seattle Gastroenterology Associates, Seattle, Washington
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Health Sciences Centre, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Mount Sinai Hospital, Toronto, Ontario